CLINICAL TRIAL: NCT02366845
Title: Prospective Validation of a Plasma Transfusion Dosing Algorithm in Patients With Chronic Liver Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-0064
Record Dates: First submitted 2015-02-04; First posted 2015-02-19 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Liver Disease
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinician Chosen Dosing (Active Comparator): Admitted University of Colorado Hospital or Denver Health bleeding patients with chronic liver disease determined to receive fresh frozen plasma (FFP) for clinical indications as determined by hospital clinician. The total dose will be determined by the physician's judgment which is the current standard of care. The physician chosen dose will be utilized but physician will be unaware of which dosing strategy has been utilized.
  INR measurements will be performed before (pre) and after (post) transfusion of plasma has been administered. Primary and secondary outcome measures will be collected. No other transfused blood component, crystalloid or colloidal fluid will be infused between the first and second INR studies except plasma.
  Interventions: Biological: Fresh Frozen Plasma; Diagnostic Test: Pre-Transfusion International Normalized Ratio (INR); Diagnostic Test: Post-Transfusion International Normalized Ratio (INR)
- Algorithm Dosing (Experimental): Admitted University of Colorado Hospital or Denver Health bleeding patients with chronic liver disease determined to receive fresh frozen plasma (FFP) for clinical indications as determined by hospital clinician. This group will receive plasma doses based on the study dosing algorithm table.
  A pre-transfusion INR (before transfusion) and a target post-transfusion INR (after transfusion) will be used to determine dose of FFP. The study table will reveal the dose in (ml/kg) of FFP to be transfused. INR measurements will be performed before (pre) and after (post) transfusion of plasma has been administered. Primary and secondary outcome measures will be collected. No other transfused blood component,crystalloid or colloidal fluid will be infused between the first and second INR studies except plasma.
  Interventions: Biological: Fresh Frozen Plasma; Diagnostic Test: Pre-Transfusion International Normalized Ratio (INR); Diagnostic Test: Post-Transfusion International Normalized Ratio (INR)

INTERVENTIONS:
Biological: Fresh Frozen Plasma — An INR dose-response curve with associated transfusion algorithm was generated for plasma in bleeding patients with chronic liver disease. In the intervention arm we will determine the plasma transfusion dose using the algorithm dosing table based on the pre-transfusion INR and the clinician chosen INR target. In the usual care group the dosing will be determined by the clinician.
  Other Names: FFP
Diagnostic Test: Pre-Transfusion International Normalized Ratio (INR) — INR result prior to Fresh Frozen Plasma (FFP) transfusion determined by clinical lab testing performed within 6 hours to 1 day before transfusion start time.
  Other Names: Pre-Transfusion INR
Diagnostic Test: Post-Transfusion International Normalized Ratio (INR) — INR result after Fresh Frozen Plasma (FFP) transfusion completed, determined by clinical lab testing performed within 1 hour after transfusion completed.
  Other Names: Post-Transfusion INR

SUMMARY:
This study plans to learn more about transfusion of a human blood component called plasma in patients who have liver problems. Patients are asked to be in this study because they have liver disease and therefore may require the transfusion of plasma.

The dose of plasma required to reach certain blood clotting laboratory targets is usually determined by clinicians. Due to the complexity of the patient's blood clotting disorder, determining the appropriate dose of plasma is very difficult. The investigators have developed a dosing table based on information from other patients with liver disease and the investigators are testing it to see if it is a more accurate dosing tool then clinician chosen dosing of plasma in patients with liver disease who need one or more plasma transfusions

DETAILED DESCRIPTION:
Clinicians currently transfuse plasma to International Normalized Ratio (INR) targets without an understanding of the dose response characteristics of plasma in bleeding patients with liver disease. Epidemiologic studies show that INR is infrequently corrected to target INR values after clinician chosen plasma transfusion doses in patients with liver disease. Plasma transfusion is frequently given to patients prior to procedures and during active bleeding in this patient population though there are no dosing guidelines to aid clinicians in reaching INR targets in patients with liver disease. Previous studies suggest that patients with liver disease may need more plasma then patients without liver disease to correct any given pre-transfusion INR (INR value measured before plasma transfusion) to the same post-transfusion INR target (INR value measured after plasma transfusion).

Current physician dosing of plasma is variable and rarely successful at reaching stated INR targets. The INR thresholds, commonly used triggers for plasma transfusion by Gastro-Intestinal (GI), Hepatology and critical care physicians at our institution range from 1.5-3.0 in bleeding or pre-procedural patients with liver disease representing tremendous variability. When we evaluated plasma transfusion dosing practices in bleeding patients with liver disease over 8 years, we demonstrated that these same physicians rarely met stated theoretical targets.

Over or under dosing plasma in these patients may lead to serious clinical complications.The target INR goal was to be within ±0.1 after the first round of FFP transfusion, and was selected because underdosing can result in prolonged bleeding, delayed procedure times, and more rounds of FFP transfusion. Furthermore, overdosing can result in excess cost, increased portal pressures, bleeding, transfusion associated circulatory overload (TACO), and transfusion related acute lung injury (TRALI).

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible to participate in the study if they meet all of the following criteria:

1. Admission to the University of Colorado Hospital or Denver Health hospital and the clinical care team plans to transfuse the patient plasma to target a specific INR value. (reason for transfusion is not considered).
2. Patient has chronic liver disease defined as 1 or more of the following: Previous diagnosis of chronic liver disease OR -Imaging or biopsy diagnosis of cirrhosis; or
3. Signs of portal hypertension (ascites, varices, hypersplenism), or
4. Laboratory evidence of synthetic dysfunction (INR>1.5, bilirubin> 2.0 mg/dL, albumin<2.5 mg/dL) AND ≥2 physical exam findings on admission associated with chronic liver disease (palmar erythema, spider angiomata, asterixis, caput medusa, gynecomastia)

Exclusion Criteria Subjects will be ineligible to participate in the study if they meet any of the following criteria

1. Patient under age 18
2. Patient actively taking vitamin K antagonists
3. Inability to obtain consent
4. Clinical team does not desire to target a specific INR value
5. Pregnant patients and prisoners
6. Patients with Acute Liver Failure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06-27 (Actual); Primary Completion 2015-06-24 (Actual); Study Completion 2019-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel C Berngard, MD, Principal Investigator — University of Colorado, Denver; Marc Moss, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

REFERENCES:
- [Background] Mannucci PM. Abnormal hemostasis tests and bleeding in chronic liver disease: are they related? No. J Thromb Haemost. 2006 Apr;4(4):721-3. doi: 10.1111/j.1538-7836.2006.01886.x. No abstract available. PMID 16634735
- [Background] Stanworth SJ, Brunskill SJ, Hyde CJ, McClelland DB, Murphy MF. Is fresh frozen plasma clinically effective? A systematic review of randomized controlled trials. Br J Haematol. 2004 Jul;126(1):139-52. doi: 10.1111/j.1365-2141.2004.04973.x. PMID 15198745
- [Background] Tripodi A. Tests of coagulation in liver disease. Clin Liver Dis. 2009 Feb;13(1):55-61. doi: 10.1016/j.cld.2008.09.002. PMID 19150309
- [Background] Iorio A, Basileo M, Marchesini E, Materazzi M, Marchesi M, Esposito A, Palazzesi GP, Pellegrini L, Pasqua BL, Rocchetti L, Silvani CM. The good use of plasma. A critical analysis of five international guidelines. Blood Transfus. 2008 Jan;6(1):18-24. doi: 10.2450/2008.0041-07. PMID 18661920
- [Background] Youssef WI, Salazar F, Dasarathy S, Beddow T, Mullen KD. Role of fresh frozen plasma infusion in correction of coagulopathy of chronic liver disease: a dual phase study. Am J Gastroenterol. 2003 Jun;98(6):1391-4. doi: 10.1111/j.1572-0241.2003.07467.x. PMID 12818286
- [Background] Sweatt AJ, Moss M, Tripputi M, Benson AB. "A dosing formula for INR-targeted plasma transfusion in bleeding patients with chronic liver disease." American Journal of Respiratory and Critical Care Medicine 2011;183:A5828
- [Background] Gajic O, Rana R, Winters JL, Yilmaz M, Mendez JL, Rickman OB, O'Byrne MM, Evenson LK, Malinchoc M, DeGoey SR, Afessa B, Hubmayr RD, Moore SB. Transfusion-related acute lung injury in the critically ill: prospective nested case-control study. Am J Respir Crit Care Med. 2007 Nov 1;176(9):886-91. doi: 10.1164/rccm.200702-271OC. Epub 2007 Jul 12. PMID 17626910
- [Background] Sorbi D, Gostout CJ, Peura D, Johnson D, Lanza F, Foutch PG, Schleck CD, Zinsmeister AR. An assessment of the management of acute bleeding varices: a multicenter prospective member-based study. Am J Gastroenterol. 2003 Nov;98(11):2424-34. doi: 10.1111/j.1572-0241.2003.t01-1-07705.x. PMID 14638344
- [Background] Maltz GS, Siegel JE, Carson JL. Hematologic management of gastrointestinal bleeding. Gastroenterol Clin North Am. 2000 Mar;29(1):169-87, vii. doi: 10.1016/s0889-8553(05)70111-4. PMID 10752021
- [Background] Benson AB, Austin GL, Berg M, McFann KK, Thomas S, Ramirez G, Rosen H, Silliman CC, Moss M. Transfusion-related acute lung injury in ICU patients admitted with gastrointestinal bleeding. Intensive Care Med. 2010 Oct;36(10):1710-1717. doi: 10.1007/s00134-010-1954-x. Epub 2010 Jul 24. PMID 20658125

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinician Chosen Dosing: University of Colorado Hospital or Denver Health bleeding inpatients with chronic liver disease receiving fresh frozen plasma (FFP) for clinical indications as determined by hospital clinician. Total dose determined by physician. (Current standard of care). Physician chosen dose will be utilized but physician blinded to which dosing strategy used.
  INR measurement performed within 1 hour after total transfusion of plasma. No other transfused blood component, crystalloid or colloidal fluid infused between the first and second INR studies except plasma
  Fresh Frozen Plasma: An INR dose-response curve with associated transfusion algorithm was generated for plasma in bleeding patients with chronic liver disease. In the intervention arm we will determine the plasma transfusion dose using the algorithm dosing table based on the pre-transfusion INR and the clinician chosen INR target. In the usual care group the dosing will be determined by the clinician.
- Algorithm Dosing: University of Colorado Hospital or Denver Health bleeding inpatients with chronic liver disease receiving fresh frozen plasma (FFP) for clinical indications as determined by hospital clinician. This group received plasma doses based on study dosing algorithm table.
  Pre-transfusion INR, target post-transfusion INR, and study table used to determine FFP dose in (ml/kg). INR measurement performed within 1 hour after entire FFP transfusion administered. No other transfused blood component,crystalloid or colloidal fluid infused between first and second INR studies except plasma.
  Fresh Frozen Plasma: An INR dose-response curve with associated transfusion algorithm was generated for plasma in bleeding patients with chronic liver disease. In the intervention arm we will determine the plasma transfusion dose using the algorithm dosing table based on the pre-transfusion INR and the clinician chosen INR target. In the usual care group the dosing will be determined by the clinician.
Period: Overall Study
Arm/Group | Clinician Chosen Dosing | Algorithm Dosing
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Clinician Chosen Dosing: Usual Care arm: Physician determined fresh frozen plasma (FFP) dosing. Bleeding patients admitted to study hospitals,with chronic liver disease determined to receive fresh frozen plasma (FFP) for clinical indications as determined by hospital clinician. Total dose determined by physician's judgment (current standard of care). Physician chosen dose will be utilized but physician will be unaware of which dosing strategy utilized.
  International Normalized Ratio (INR) measurement will be performed within 1 hour after entire plasma transfusion administered. No other transfused blood component, crystalloid or colloidal fluid infused between first and second INR studies except plasma.
- Algorithm Dosing: Intervention arm: Plasma transfusion dose determined using algorithm dosing table based on the (pre-transfusion INR) and clinician chosen INR target. Bleeding patients admitted to study hospitals with chronic liver disease determined to receive fresh frozen plasma (FFP) for clinical indications as determined by hospital clinician.
  Pre-transfusion INR and target post-transfusion INR used to determine FFP dose. The study table determines dose in (ml/kg) of FFP. INR measurement will be performed within 1 hour after entire plasma transfusion administered. No other transfused blood component,crystalloid or colloidal fluid will be infused between the first and second INR studies except plasma.
- Total: Total of all reporting groups
Arm/Group | Clinician Chosen Dosing | Algorithm Dosing | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (11.1) | 53.3 (10.7) | 53.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 15 | 16 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 13 | 16 | 29
  Black or African American | 2 | 1 | 3
  Hispanic or Latino | 9 | 8 | 17
  Asian | 0 | 1 | 1
Pre-Transfusion International Normalzied Ratio (INR) [Mean (Standard Deviation); unit: ratio] — International Normalized Ratio (INR) laboratory blood value measured before start of plasma transfusion. Laboratory tests performed within 1 day were acceptable, if the values were stable for the proceeding 2 days and there was no change in patient's clinical status. Otherwise, a pre-transfusion INR was obtained within 6 hours of transfusion start time.
  ratio | 2.4 (0.5) | 2.3 (0.4) | 2.3 (0.5)
Physician target International Normalized Ratio (INR) [Mean (Standard Deviation); unit: ratio] — Prior to randomization, the treating clinical physician who was responsible for making the plasma dosing decision identified their desired INR target.
  ratio | 1.7 (0.2) | 1.8 (0.2) | 1.7 (0.2)
Hospital Service [Number; unit: participants]
  Medical Floor | 23 | 22 | 45
  Other | 1 | 4 | 5
Serum Creatinine [Geometric Mean (Inter-Quartile Range); unit: mg/dL] | 1.3 [1.0 to 1.8] | 1.2 [1.0 to 1.5] | 1.3 [1.1 to 1.5]
APACHE II Score [Mean (Standard Deviation); unit: units on a scale] — APACHE II (Acute Physiology And Chronic Health Evaluation II) is a severity-of-disease classification system with a final score of 0 to 71. Higher scores correspond to more severe disease and higher risk of death.
  The weighted score uses 12 of the most commonly measured physiologic measures in hospitalized patients: vital signs (heart rate, mean blood pressure, respiratory rate, temperature and Glasgow Coma Score), routine blood test values (hematocrit and white blood cell count, serum potassium, serum sodium, serum creatinine), and arterial blood gas values (serum pH and Pa02).
  units on a scale | 13.9 (6.7) | 13.9 (3.5) | 13.9 (5.3)
MELD Score [Mean (Standard Deviation); unit: units on a scale] — The Model of End-stage Liver Disease (MELD) Score is a validated scoring system to estimate relative disease severity and likely survival of patients awaiting liver transplantation.
  Score range is 6 to 40, with higher scores corresponding to more severe disease. Weighted patient laboratory values for serum bilirubin, serum creatinine, and the international normalized ratio (INR) for prothrombin time predict three-month survival. In patients with cirrhosis, an increasing MELD score is associated with increasing severity of hepatic dysfunction and increased three-month mortality risk.
  units on a scale | 25.9 (8.4) | 25.4 (5.4) | 25.6 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Reached Targeted International Normalized Ratio (INR) Within ±0.1 After First Fresh Frozen Plasma (FFP) Transfusion Completed.
Description: Ability of dosing algorithm to accurately predict necessary plasma dose (ml/kg), required to reach commonly targeted International Normalized Ratio (INR) values, compared to clinician chosen plasma transfusion dose, as determined by dose-response curve.
  The primary outcome was achievement of the target INR within ±0.1 after the first round of FFP transfusion. This primary outcome was selected because underdosing can result in prolonged bleeding, delayed procedure times, and more rounds of FFP transfusion. Furthermore, overdosing can result in excess cost, increased portal pressures, bleeding, transfusion associated circulatory overload (TACO), and transfusion related acute lung injury (TRALI).
Time Frame: within 1 hour after entire plasma transfusion
Population: At goal INR after first transfusion.
Measure: Count of Participants; unit: Participants
Groups:
- Clinician Chosen Dosing: Usual Care arm: Physician determined FFP dosing. Bleeding patients admitted to study hospitals,with chronic liver disease determined to receive fresh frozen plasma (FFP) for clinical indications as determined by hospital clinician. Total dose determined by physician's judgment (current standard of care). Physician chosen dose will be utilized but physician will be unaware of which dosing strategy utilized.
  INR measurement will be performed within 1 hour after entire plasma transfusion administered. No other transfused blood component, crystalloid or colloidal fluid infused between first and second INR studies except plasma
- Algorithm Dosing: Intervention arm: Plasma transfusion dose determined using algorithm dosing table based on the pre-transfusion INR and clinician chosen INR target. Bleeding patients admitted to study hospitals with chronic liver disease determined to receive fresh frozen plasma (FFP) for clinical indications as determined by hospital clinician.
  Pre-transfusion INR and target post-transfusion INR used to determine FFP dose. The study table determines dose in (ml/kg) of FFP. INR measurement will be performed within 1 hour after entire plasma transfusion administered. No other transfused blood component,crystalloid or colloidal fluid will be infused between the first and second INR studies except plasma.
Arm/Group | Clinician Chosen Dosing | Algorithm Dosing
Number analyzed (Participants) | 24 | 26
Participants | 7 | 17

2. Secondary Outcome: Time (Hours) From Initiation of First Dose of Plasma to Initiation of Planned Procedure (in Patient Undergoing Transfusion Before a Procedure) for Clinician Dosing Compared to Algorithm Dosing Strategies.
Description: Decreased time between initiation of plasma infusion, achieving a corrected target INR and start of planned patient procedures would potentially improve care efficiency and/or allow faster intervention in unstable patients.
Time Frame: hours from first dose to initiation of procedure, anticipated timeframe between 1 minute to 8 hours.
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Clinician Chosen Dosing | Algorithm Dosing
Number analyzed (Participants) | 24 | 26
hours | 4.9 [3.5 to 6.8] | 3.5 [2.7 to 4.5]

3. Secondary Outcome: Dose Difference (Average # Units) Between Clinician Dosing and Algorithm Dosing (Units of FFP) Per Patient.
Time Frame: within 1 hour after entire plasma transfusion
Measure: Mean (95% Confidence Interval); unit: units
Arm/Group | Clinician Chosen Dosing | Algorithm Dosing
Number analyzed (Participants) | 24 | 26
units | 2.4 [1.9 to 3.0] | 3.1 [2.5 to 3.9]

4. Secondary Outcome: Hospital Length of Stay
Time Frame: Subjects will be followed for duration of hospital stay, anticipated within 1 Day to 28 Days
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Clinician Chosen Dosing | Algorithm Dosing
Number analyzed (Participants) | 24 | 26
days | 13.8 [9.8 to 19.4] | 11.0 [7.0 to 17.2]

ADVERSE EVENTS:
Arm/Group | Clinician Chosen Dosing | Algorithm Dosing
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No